CLINICAL TRIAL: NCT03417869
Title: QuickVue Influenza A + B Test Field Study
Acronym: QuickVue Flu
Status: Completed | Type: Observational
Sponsor: Quidel Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-0103-02
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Influenza A, Influenza B

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: QuickVue Influenza A+B — Rapid diagnostic test with IVD, QuickVue Influenza A+B

SUMMARY:
Demonstrate improved clinical performance of visually read QuickVue Influenza A+B test.

DETAILED DESCRIPTION:
The objective of this study is to demonstrate an improved clinical performance of the visually read QuickVue Influenza A+B test with nasal and nasopharyngeal swab specimens. Clinical performance will be based on comparison of QuickVue results to either cell culture or an FDA-cleared molecular test at one or more Reference Laboratories.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be recruited from the general population as they present to the clinical facility. Subjects must have had a fever within the last two days and exhibiting one or more symptoms characteristic of influenza. They must meet the following criteria to be eligible for enrollment:

1. Male or Female of all ages (with appropriate consent).
2. The subject must have had of a fever, ≥ 37.8º C (100º F), within the last two days.
3. Must also be currently exhibiting one or more of the following symptoms characteristic of influenza-like-illness (ILI).

   1. Nasal congestion
   2. Rhinorrhea
   3. Sore throat
   4. Cough
   5. Headache
   6. Myalgia
   7. Malaise

Exclusion Criteria:

* 1. Has undergone treatment with anti-influenza antivirals within the previous 7 days, to include but not be limited to, Amantadine, Rimantadine, Ribavirin, Oseltamivir, Zanamivir or any other antiviral currently available in these classes.

  2. Has been vaccinated by means of an influenza nasal spray/mist vaccine within the previous 7 days.

  3. Unable to understand and consent to participation; for minors this includes parent or legal guardian.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited from the general population as they present to the clinical facility. Subjects must have had a fever within the last two days and exhibiting one or more symptoms characteristic of influenza
Sampling Method: Probability Sample
Enrollment: 1381 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Influenza Diagnostic test result | 10 minutes
  rapid IVD test

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Alliance Urgent Care, Phoenix, Arizona
  - Twelve Corners Pediatrics, Rochester, New York
  - Veritas, P.A., Belton, Texas
  - City Doc Urgent Care, Dallas, Texas
  - Advanced Pediatrics, Vienna, Virginia

IPD SHARING:
Plan to Share IPD: No